CLINICAL TRIAL: NCT00960921
Title: Study of the Effects of Iron Supplementation on High Altitude Pulmonary Hypertension.
Brief Title: Study of the Effects of Iron on Lung Blood Pressure at High Altitude
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started.
Sponsor: University of Oxford (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oxford-Kyrgyzstan-2009
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary artery pressure; Hypoxia; Iron; Hypoxia-inducible factor; High altitude
MeSH Terms: conditions — Hypertension, Pulmonary; Hypoxia; Altitude Sickness | interventions — Ferric Oxide, Saccharated; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron group (Experimental): Patients with high altitude pulmonary hypertension receive six intravenous infusions of iron sucrose, administered on days 0, 4, 8, 12, 16 and 20 of the study. The total study period is 28 days. Pulmonary artery systolic pressure is measured before each infusion, and again on day 28.
  Interventions: Drug: Iron sucrose
- Saline group (Placebo Comparator): Patients with high altitude pulmonary hypertension receive six intravenous infusions of normal saline, administered on days 0, 4, 8, 12, 16 and 20 of the study. The total study period is 28 days. Pulmonary artery systolic pressure is measured before each infusion, and again on day 28.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Iron sucrose — An intravenous infusion of 100 mg of iron is administered on days 0, 4, 8, 12, 16 and 20 of the study, giving a total of six iron infusions for each participant in the iron group over the course of the 28-day study period.
  Other Names: Venofer (iron sucrose)
  Arms: Iron group
Drug: Normal saline — An intravenous infusion of 100 ml of normal (0.9 %) saline is administered on days 0, 4, 8, 12, 16 and 20 of the study, giving a total of six saline (placebo) infusions for each participant in the saline group over the course of the 28-day study period.
  Arms: Saline group

SUMMARY:
Body iron levels may be important in determining how the blood pressure in the lungs changes in response to low oxygen levels. At high altitude, where oxygen levels are low, some patients develop elevated lung blood pressure. The investigators hypothesize that, in high altitude residents with elevated lung blood pressure, iron supplementation will cause a reduction in lung blood pressure.

DETAILED DESCRIPTION:
Pulmonary hypertensive disorders frequently complicate hypoxic lung disease and worsen patient survival.

Hypoxia-induced pulmonary hypertension is also a major cause of morbidity at high altitude. Hypoxia causes pulmonary hypertension through hypoxic pulmonary vasoconstriction and vascular remodelling. These processes are thought to be regulated at least in part by the hypoxia-inducible factor (HIF) family of transcription factors, which coordinate intracellular responses to hypoxia throughout the body.

HIF is regulated through a cellular degradation process that requires iron as an obligate cofactor. In cultured cells HIF degradation is inhibited by reduced iron availability (by chelation with desferrioxamine) and potentiated by iron supplementation. In humans, laboratory experiments lasting eight hours have shown that acute iron supplementation blunts the pulmonary vascular response to hypoxia, while acute iron chelation with desferrioxamine enhances the response.

These findings suggest that iron may also affect the pulmonary vascular response to hypoxia over longer time periods. The purpose of this study, which will take place at high altitude in Kyrgyzstan, is to investigate whether iron supplementation can reduce pulmonary artery pressure in patients with established high altitude pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* High altitude natives, currently resident at high altitude
* Pulmonary hypertension (mean pulmonary artery pressure > 25 mmHg)
* Pulmonary artery systolic pressure measurable using Doppler echocardiography

Exclusion Criteria:

* Clinical evidence or history of major co-morbidity
* Recent changes to relevant medications, or taking iron/vitamin supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary artery systolic pressure | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Robbins, DPhil BM BCh, Principal Investigator — University of Oxford
Locations (1):
- Institute of Molecular Biology and Medicine, Bishkek, Kyrgyzstan